CLINICAL TRIAL: NCT00738686
Title: Austrian Multivessel Taxus-Stent Registry
Acronym: AUTAX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Helmut-Dietmar Glogar, Dept. Cardiology, Medical University of Vienna, Austria
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUTAX
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; drug-eluting stent; percutaneous coronary intervention; major adverse cardiac event; in-stent restenosis; stent thrombosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Single-arm study, no placebo or control group
  Interventions: Device: Intracoronary stent implantation

INTERVENTIONS:
Device: Intracoronary stent implantation — Taxus stent implantation in patients with multivessel coronary artery disease
  Other Names: Taxus Express; Taxus Liberte

SUMMARY:
The aim of AUTAX study is to investigate the frequency of MACCE in patients with multivessel disease and multiple Taxus stent implantations in the "real world" stenting at 30 days, 6 and 12 months at 2 year follow-up. Because multivessel stenting using DES has been limited due to economic considerations, the secondary aim is to enhance experience in multivessel stenting with drug-eluting stents in order to improve short- and long-term outcomes of the patients with severe multiple coronary artery stenoses.

The objectives of the study are:

1. To determine the frequency of MACCE at 30-day, 6 and 12-month and at 2 year clinical follow-up after multivessel intervention with drug-eluting stents in a prospective patient cohort..
2. To determine the rate of in-stent restenosis, target lesion and target vessel revascularization (angiographic measures) 6 months in patients with multiple DESs in multiple lesions.
3. To investigate the clinical and angiographic outcomes after implantation of multiple DESs in the subgroup of patients with accompanying diseases (diabetes mellitus, renal insufficiency) with known high restenosis and late complication rate.
4. To evaluate potential cost burden in attempting a strategy of complete revascularization by multiple DES in patients with multivessel disease.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic coronary multivessel disease
* possible percutaneous complete coronary revascularization
* age >18 year
* significant coronary lesion at least in 2 vessels

Exclusion Criteria:

* acute myocardial infarction within 48 hours
* contraindications to clopidogrel, aspirin, heparin and taxol
* pregnancy or lack of protection against pregnancy or breast-feeding during the study
* hemorrhagic diathesis
* platelet count <100.000/ml3

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2004-06; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Incidence of MACCE, defined as all-cause death, nonfatal acute myocardial infarction (AMI) target vessel revascularization (TVR) and cerebrovascular event during the two-year clinical follow-up (FUP) | 2 year

SECONDARY OUTCOMES:
Break-down primary endpoints at the 2-year FUP, as the rate of TVR, non-fatal AMI, all-cause death, stroke and the composite of death and AMI | 2 year
Incidence of 30-days, 6-mo and 1-year MACCE | 1 year
Acute, subacute and late thrombosis rates | 2 year
Angiographic end-points as the binary restenosis rate per lesion (defined as diameters stenosis ≥ 50%), in-stent and proximal and distal in-lesion late lumen loss | 6-month

CONTACTS AND LOCATIONS:
Overall Officials: Helmut-Dietmar Glogar, MD FESC, Principal Investigator — Dept. Cardiology, Medical University of Vienna, Vienna, Austria
Locations (7):
- Austria (7):
  - Landeskrankenhaus, Bruck an der Mur
  - Department of Interventional Cardiology, Academic Hospital, Feldkirch
  - Landeskrankenhaus Graz-West, Graz
  - Allgemeines Krankenhaus der Stadt Linz, Linz
  - Krankenhaus Barmherzigen Schwestern, Linz
  - St. Johannes Spital, Salzburg
  - Rudolfstiftung, Vienna

REFERENCES:
- [Derived] Gyongyosi M, Christ G, Lang I, Kreiner G, Sochor H, Probst P, Neunteufl T, Badr-Eslam R, Winkler S, Nyolczas N, Posa A, Leisch F, Karnik R, Siostrzonek P, Harb S, Heigert M, Zenker G, Benzer W, Bonner G, Kaider A, Glogar D; AUTAX Investigators. 2-year results of the AUTAX (Austrian Multivessel TAXUS-Stent) registry beyond the SYNTAX (synergy between percutaneous coronary intervention with TAXUS and cardiac surgery) study. JACC Cardiovasc Interv. 2009 Aug;2(8):718-27. doi: 10.1016/j.jcin.2009.05.019. PMID 19695539